CLINICAL TRIAL: NCT04233788
Title: Metabolic Characterization of Space Occupying Lesions of the Brain Using in Vivo MR- (Spectroscopic) Imaging at 3 Tesla and 7 Tesla
Brief Title: Metabolic Characterization of Space Occupying Lesions of the Brain
Acronym: FASTMRSI
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00503
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Brain Tumor; Glioma; IDH Mutation
Keywords: Magnetic Resonance Spectroscopic Imaging (MRSI); Chemical exchange saturation transfer imaging (CEST); Pulse sequence development; Preoperative prediction of IDH-status; Quantitative MR(S)I; Signal processing
MeSH Terms: conditions — Brain Neoplasms; Glioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Sequence optimization (Healthy Control Group 1 (10 Persons)): The MEGA-based editing sequences as well as the SLOW-EPSI sequence will be applied to this group using a 3T Prisma and a 7T Terra scanner. Data will be used for optimization of the pulse sequences.
  Aim: find those sequence parameters to obtain best spectral quality data (SNR, spatial resolution versus measurement time).
  Interventions: Device: MR-scans using a 3T Prisma and a 7T Terra scanner (Siemens, Erlangen Germany)
- Healthy Control Group 2 (15 Persons): The best performing sequence which will be applied to this group using a 7T Terra scanner. Data will be used normative data for glutamate/glutamine and GABA levels in healthy controls.
  Aim: normal reference data for future studies.
  Interventions: Device: MR-scans using a 3T Prisma and a 7T Terra scanner (Siemens, Erlangen Germany)
- Patient Group 1: Comparison of 5 different spectral editing sequences (30 Patients): Two editing pulse sequence types will be applied to this group at a 3T Prisma and a 7T Terra scanner. The sequences being compared are MEGA-semiLASER-SVS, MEGA-semiLASER based MRSI (on both 3T and 7T) and SLOW-EPSI (on 7T only).
  Interventions: Device: MR-scans using a 3T Prisma and a 7T Terra scanner (Siemens, Erlangen Germany)
- Patient Group 1: Comparison of 4 different CEST sequences (30 Patients): Two different CEST sequence types will be applied to this group at a 3T Prisma and a 7T Terra scanner. The CEST performance will be compared between 3T and 7T, as well which of the two types in the best on each scanner.
  Aim: which of the four sequence predicts the IDH-mutation status best.
  Interventions: Device: MR-scans using a 3T Prisma and a 7T Terra scanner (Siemens, Erlangen Germany)

INTERVENTIONS:
Device: MR-scans using a 3T Prisma and a 7T Terra scanner (Siemens, Erlangen Germany) — The MR-scans performed at 3T and 7T are performed to evaluate whether high field MR-examinations bring an advantage to the patient in determining the IDH-status of the glioma. Two MRSI/CEST sequences will be tested against each other.
  Other Names: Examined are fast MRSI sequences and CEST sequences.

SUMMARY:
High field MR-technologies are expected to boost metabolic spectroscopic imaging (MRSI), but also CEST-MRI. This is due to the fact that increased SNR is available which can be used to increase the spatial resolution of all sequences, or reduction of measurement times. Recent findings has shown that MRSI can be used to evaluate the isocitrate dehydrogenase (IDH) status of gliomas, a brain tumor type which is most often diagnosed in humans. Patients with IDH-mutated gliomas have a much longer survival time that IDH-wildtype. In IDH-mutated gliomas the substance 2-hydroxy-glutarate (2HG) is found, whereas in IDH-wildtype gliomas it is not.

The underlying trial aims to measure 2HG directly with different MRSI sequences at 3 Tesla (3T) and 7 Tesla (7T) magnetic field strength. Apart from MRSI-techniques for IDH-typing it has been shown that CEST-imaging can also be performed to determine the IDH-status of gliomas.

A total of 75 patients and 50 healthy controls will be examined in this study to evaluate the most accurate method for pre-operative IDH-status determination.

DETAILED DESCRIPTION:
Introduction - Recently the first commercially available 7T MR-scanner which is approved for clinical use came on to the market. The main motivation to go to higher field strengths is the fact that better SNR can be achieved in shorter acquisition time, or higher spatial resolution can be obtained in the same measurement time. High field MRI also has drawbacks, e.g. substantially higher specific absorption rate (SAR), higher susceptibility related image distortion problems, and longer longitudinal relaxation times. Nevertheless, moving to higher fields is especially beneficial for MR-spectroscopy. This is due to the fact that better signal to noise ration (SNR) is combined with higher spectral resolution. The two most commonly used techniques for spectroscopic imaging (MRSI) are: (i.) relative slow 2D/3D techniques like PRESS and semiLASER based techniques, and (ii.) fast 3D echo planar based (EPI) techniques. Although echo planar spectroscopic imaging (EPSI) is a technique that has been introduced by Sir Peter Mansfield in the first half of 80es, the method is still continuously being improved, and recently very promising applications related to brain tumor diagnostics were published. To be mentioned in this context is the fact that the method can be combined with spectral editing for the detection of 2-hydroxy-glutarate (2HG) in glioma patients. 2HG is only present if the glioma that has mutations in the IDH-gene. It is shown that gliomas having the IDH-mutation have a much better overall survival prognosis. Apart from brain tumor typing, high resolution EPSI imaging also enables investigation the investigation of tumor infiltration using metabolic criteria. In surgery the patients' preoperative intake of the 5-aminolevulinic acid (5-ALA) before surgery selectively makes malignant glioma tissues fluorescent under blue light irradiation and tumor itself becomes clearly visible during the neurosurgical intervention. The fact that 5-ALA-guided completely-resected glioma patients have a significant longer survival time, underlines the necessity to know the exact tumor boundaries.

Aims - The major aims of the study proposed are manifold:

(i.) The development of a novel EPSI-pulse sequence utilizing 3D-radial k-space sampling schemes, that focuses on robustness w.r.t. patient motion, is robust with respect to chemical shift displacement artifacts, includes the possibility of 2HG-spectral editing, uses SAR-reduced radiofrequency (RF) pulses, and operate with total acquisition times that are acceptable for clinical routine use; (ii.) Comparison of the novel sequence with available conventional EPSI-techniques and semiLASER-based techniques for clinical routine use comparing its performance at 3T and 7T; (iii.) The development of a graphic processor unit (GPU) based fitting algorithm for quantification of 3D-radial EPSI-data based on the existing tdfdfit-algorithm; (iv.) Extension of a locally developed machine learning based automatic quality-filtering algorithm to be applied on the researchers' novel EPSI-data; (v.) Quantitative investigation on the effect spatial non-uniform transmit and receive properties for all relevant metabolites and spatial dependent signal amplitude correction schemes (extension of a locally developed method); (vi.) Investigation of the exact effects of selective excitation on J-coupled spin systems, and comparison of these effects between 3T and 7T; (vii.) Reproducibility study on 20 healthy volunteers measured twice with the same protocol (10 recorded twice at 7T and 10 recorded twice at 3T); (viii.) Pre-operative application of the best suited EPSI-pulse sequence in a total of 75 patients. All patients will be recorded at 3T as well as at 7T using the equivalent protocols; (ix.) Co-registration of pre-operative, spatially resolved 3D-EPSI-MRSI data with post-operative 3D-FLAIR and T1c-imaging in IDH-wildtype patients with had complete resection during 5-ALA guided neurosurgical interventions will provide information on whether MRSI-techniques are helpful to predict the tumor affected volume; (x.) Documentation of the location of a biopsy, histology to enable a better correlation between MR-spectroscopic patterns and histology.

(xi) Comparison of the performance of CEST versus the CMRR-semiLASER MRSI sequence w.r.t. to the prediction accuracy of the IDH-type of the glioma by the two technologies.

Methodology - The implementation of a robust EPSI sequence that uses 3D-radial k-space sampling schemes and reconstruction will be performed on Siemens IDEA developer platforms for VE- and XA-software versions. The sequence will be compared to the performance obtained with another EPSI implementation, available via Siemens, as well as the CMRR-implementation of the MEGA (MEscher-GArwood) semi-LASER (Localization by Adiabatic SElective Refocusing) for 2HG-editing (CMRR Spectroscopy Package, 2012). The quantification of the EPSI-data of the reference sequence will be performed with the MIDAS package. The EPSI-data of the novel sequence as well as MEGA-semi-LASER sequence will be quantified using a parallelized GPU-re-implementation of the tdfdfit-algorithm made available as separate plugin within jMRUI-spectroscopy package (jMRUI: java magnetic resonance user interface). Co-registration of pre-surgery EPSI-data with post-operative structural MRI-data will be performed with the SPM (Statistical Parameter Mapping) program. Further statistical analysis and machine learning algorithms will be based on statistical programming language "R". The CEST pulse sequences will be obtained via Siemens-Healthineers.

Potential significance - (a.) Pre-surgical knowledge of the IDH-status will enable better individual neurosurgical treatment of the patient; (b.) Coregistration of metabolic EPSI-data, with post-operative structural MR-data will give information on the fundamental usefulness of MRSI-techniques to detect glioma infiltration zones; (c.) Improved follow-up of IDH-mutated glioma patients, who typically have a long period of minimal progression, followed rapidly by aggressive growth and transformation to higher grade; (d.) The availability of an imaging biomarker to monitor tumor recurrence would be a major advance for all glioma patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people who are able to lie in the MR scanner for one hour;
* Patients with suspected mass in the brain
* Written informed consent

Exclusion Criteria:

* Persons under the age of 18
* Persons who are mentally unable to choose to participate
* Pregnant women
* Patients with oncological findings or neurodegenerative findings in the past
* Wearing active implants (e.g. pacemakers and neurostimulators)
* Emergency patients
* Persons with tattoos on the head or neck area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls: Each of the participating healthy adult persons in the study will receive 2 out of 5 different pulse sequences which will be tested against each other (5 groups with 10 healthy controls). In each group two pulse sequences will be tested against each other at 3T and 7T. The data of the healthy controls will be used an normal values to compare patient data against.
  Patients: 75 patients will be also be split in 5 groups groups of 15 patients. Each patient will receive 2 out of 5 MRSI and/or CEST pulse sequences which will be tested against each other in that group. The best pulse sequence is propagated to the next group. The pulse sequences will be applied at 3T and at 7T (when available). With this approach the researchers hope to find out the most accurate sequence that predicts the IDH-status pre-operatively.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Optimal MR-sequence for IDH-typing | 48 months
  Finding the most optimal (2HG-edited, radial kspace-sampled) EPSI MRSI/CEST technique for the initial diagnosis of gliomas with respect to IDH-typing. Pre-operative knowledge of the IDH-type is important information for further neurosurgical treatment.

SECONDARY OUTCOMES:
Spectral/CEST pattern | 48 months
  The retrospective analysis of tumor affected tissue volumes identified by 3D-MRSI/CEST image data with the factual resected volumes during 5-ALA guided complete tumor resection interventions enable to find the relationship between the spectral or CEST pattern and the location of the glioma.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Slotboom, PhD, Study Chair — University of Bern
Locations (1):
- Institute for Diagnostic and Interventional Neuroradiology, University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paech D, Windschuh J, Oberhollenzer J, Dreher C, Sahm F, Meissner JE, Goerke S, Schuenke P, Zaiss M, Regnery S, Bickelhaupt S, Baumer P, Bendszus M, Wick W, Unterberg A, Bachert P, Ladd ME, Schlemmer HP, Radbruch A. Assessing the predictability of IDH mutation and MGMT methylation status in glioma patients using relaxation-compensated multipool CEST MRI at 7.0 T. Neuro Oncol. 2018 Nov 12;20(12):1661-1671. doi: 10.1093/neuonc/noy073. PMID 29733378
- [Background] Choi C, Ganji SK, DeBerardinis RJ, Hatanpaa KJ, Rakheja D, Kovacs Z, Yang XL, Mashimo T, Raisanen JM, Marin-Valencia I, Pascual JM, Madden CJ, Mickey BE, Malloy CR, Bachoo RM, Maher EA. 2-hydroxyglutarate detection by magnetic resonance spectroscopy in IDH-mutated patients with gliomas. Nat Med. 2012 Jan 26;18(4):624-9. doi: 10.1038/nm.2682. PMID 22281806
- [Background] Marjanska M, Auerbach EJ, Valabregue R, Van de Moortele PF, Adriany G, Garwood M. Localized 1H NMR spectroscopy in different regions of human brain in vivo at 7 T: T2 relaxation times and concentrations of cerebral metabolites. NMR Biomed. 2012 Feb;25(2):332-9. doi: 10.1002/nbm.1754. Epub 2011 Jul 27. PMID 21796710
- [Background] Sabati M, Sheriff S, Gu M, Wei J, Zhu H, Barker PB, Spielman DM, Alger JR, Maudsley AA. Multivendor implementation and comparison of volumetric whole-brain echo-planar MR spectroscopic imaging. Magn Reson Med. 2015 Nov;74(5):1209-20. doi: 10.1002/mrm.25510. Epub 2014 Oct 29. PMID 25354190
- [Background] Slotboom J, Boesch C, Kreis R. Versatile frequency domain fitting using time domain models and prior knowledge. Magn Reson Med. 1998 Jun;39(6):899-911. doi: 10.1002/mrm.1910390607. PMID 9621913